CLINICAL TRIAL: NCT04216498
Title: Describing Relationships Between Psychosocial Outcomes and Readiness for Transition in Adolescent and Young Adult Patients With Juvenile Idiopathic Arthritis - a Pilot Study
Brief Title: Psychosocial Outcomes and Transition Readiness in JIA
Status: Completed | Type: Observational
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Collaborators: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: SCH-2109
Record Dates: First submitted 2018-05-21; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pre-Transfer Patients aged 10-16 years
- Post-Transfer Patients aged 16-25 years
- Parents/Guardians of Pre-Transfer Patients

SUMMARY:
It is widely acknowledged that the transition from paediatric to adult health services should be a multidimensional and multidisciplinary process that addresses the medical, psychosocial, and educational needs of adolescents and young adults (AYA). Despite this, there is currently a scarcity of research examining the relationships between psychosocial factors (e.g., anxiety, social support) and transition readiness in AYA with juvenile idiopathic arthritis (JIA). This study therefore aimed to examine the relationships between psychosocial factors and transition readiness in pre-transfer adolescents and post-transfer young adults aged 10-25 years diagnosed with JIA at a single centre.

In total, 40 adolescents aged 10-16 years together with a parent/guardian, will take part at Sheffield Children's Hospital and 40 young adults aged 16-25 years will take part at Sheffield Teaching Hospitals. Participants will be asked to complete a battery of self-report questionnaire measuring psychosocial factors (anxiety/depression, social support, family functioning, health-related quality of life) and transition readiness (transition knowledge and skills, self-efficacy). JIA disease severity was also measured during clinic appointments. This study has received full ethical approval, and all participants will give their written informed assent or consent before taking part.

The results from this research will be important in better understanding which psychosocial factors affect how ready young people with JIA feel to move from paediatric to adult rheumatology services. We hope this research will inform further work to help target psychological interventions in this group of patients.

ELIGIBILITY:
Patient Inclusion Criteria:

* Aged 10-25 years
* Diagnosis of juvenile idiopathic arthritis (including all ILAR subtypes except 'systemic arthritis' and 'undifferentiated arthritis')
* Juvenile idiopathic arthritis managed by Sheffield Children's Hospital or Sheffield Teaching Hospitals
* Fluent in verbal and written English

Patient Exclusion Criteria:

* Aged <10 years or >25 years
* Diagnosis of juvenile idiopathic arthritis ILAR subtypes 'systemic arthritis' or 'undifferentiated arthritis')
* Diagnosis of uveitis
* Non-fluent in verbal and written English

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will be patients aged 10-25 years or parents/guardians of patients aged 10-16 years who have a diagnosis of juvenile idiopathic arthritis.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Generalised Anxiety | 1 day
  Generalised Anxiety Disorder-7 Questionnaire (Spitzer et al., 2006)

SECONDARY OUTCOMES:
Depression | 1 day
  Patient Health Questionnaire-9 Questionnaire (Spitzer et al., 1999)
Health-related quality of life | 1 day
  Paediatric Quality of Life Arthritis Module (Varni et al., 2002)
Social support | 1 day
  Bath Adolescent Pain Questionnaire Social Support Subscale (Eccleston et al., 2005)
Family functioning | 1 day
  Bath Adolescent Pain Questionnaire Family Functioning Subscale (Eccleston et al., 2005)
Prosocial and problem behaviours | 1 day
  Strengths and Difficulties Questionnaire (Goodman, 1997)
JIA disease severity (JADAS-3) | 1 day
  JADAS-3 is a composite score of patient VAS score, physician VAS score, active joint count

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Children's NHS Foundation Trust, Sheffield, United Kingdom